CLINICAL TRIAL: NCT04214223
Title: Validation of a New Tool for a Numeric Pre-anesthesic Evaluation for Pregnant Women During Their Pregnancy Follow-up in University and Regional Maternity of Nancy (France)
Brief Title: Conception of a Decisional Tool Using a Pre-Anesthesic Numerical Evaluation (PANE) During the 8th Month of Pregnancy
Acronym: PANE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI140
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy Related
Keywords: Pregnancy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PANE -> PAC: First, the patient carry out her Pre-Anesthesic Numerical Evaluation and then she benefits from her Pre-Anesthesic Consultation.
  Interventions: Other: Pre-Anesthesic Consultation; Other: Pre-Anesthesic Numerical Evaluation
- PAC -> PANE: First, the patient benefits from her Pre-Anesthesic Consultation and then, she carry out her Pre-Anesthesic Numerical Evaluation
  Interventions: Other: Pre-Anesthesic Consultation; Other: Pre-Anesthesic Numerical Evaluation

INTERVENTIONS:
Other: Pre-Anesthesic Consultation — Classical Pre-Anesthesic Consultation with an anesthesist of the maternity hospital of Nancy (France)
Other: Pre-Anesthesic Numerical Evaluation — Home-based Pre-Anesthesic Numerical Evaluation with the aid of a questionnaire, achieved with a computer, digital tablet or smartphone, on a secured platform.

SUMMARY:
In France, all pregnant women benefit from an pre-anesthesic consultation (PAC) to evaluate their physical and biological conditions.

Many of pregnant women are healthy, there is only on type of induction protocol in case of general anesthesia, they are all at risk of difficult intubation and blood samples are already performed by obstetricians.

Thus, investigators' hypothesis is that for many pregnant women, an alternative pre-anesthesic evaluation, other than the classic 8th month PAC is possible. So, the investigators would create a tool able to perform a women's triage, and to detect which of them have to see an anesthesist during a face-to-face consultation and which of them could do without it.

Investigators' study will be about the monocentric analysis of a pre-anesthesic numerical evaluation with the aid of a questionnaire, vouched for by an experts committee specialized in obstetrical anesthesia.

DETAILED DESCRIPTION:
Every month, several thousands of women benefit from an obstetrical pre-anesthesic consultation (PAC) in France, during their 8th month of pregnancy. It is the opportunity to evaluate women's physical and biological conditions before their delivery.

This consultation is mandatory in France. It must be carried out by an anesthesist and should aim at proposing an analgesic and anesthesic strategies as well as relaying all the resulting information to the patients.

A study carried out in 2015 in two Parisian 3rd level maternity hospitals showed that the majority of women seen in obstetrical PAC are healthy. A preliminary observational, prospective and multicentric study in 20 Lorraine (France) maternity hospitals was implemented in order to identify more specifically the population of women seen during this consultation. Despite of a probable under-estimation, investigators' results showed 40,3% of women ASA 1, with a physiologic pregnancy, without hemostasis disorder and planned for a vaginal delivery.

With these healthy women, according to the recommendations of the French Society of Anesthesia and Intensive Care (SFAR) edited in 2012 and those of the French Health Authority (HAS) edited in 2016, the only obligatory biological exam for the anesthesic care is the 6th month blood count (with blood type and irregular antibodies).

Despite those recommendations, over-prescription of biological tests during the preoperative clinic in pre-partum persists (in the investigators' study, they found a probable under-estimated number of 34,5% unjustified prescriptions).

Moreover, the PAC aims at evaluating superior airways, for the purpose of a potential oro-tracheal cannulation in case of general anesthesia. However, this evaluation had a relative interest in this context considering that the superior airways anatomy changes during pregnancy and labor and all pregnant women must all be considered at risk of difficult intubation.

In addition, all pregnant women from 20 weeks of amenorrhea are considered as full stomach. Thus, in case of general anesthesia, the investigators have to perform a crash induction. So, there is no other protocol of induction to consider in this context.

Regardless of the context, pregnant women see an anesthesist before their delivery during the pre-anesthesic visit : the sooner 24 hours before an intervention, at the latest when they arrive in the delivery room.

Actually, society is faced with important problems of medical demography and anesthesists are less and less numerous, making their activity more and more difficult.

Investigators' hypothesis is that for the population of pregnant healthy women, an alternative pre-anesthesic evaluation, other than the classic 8th month PAC, could be an innovative idea for health system, ensuring care quality and security of pregnant women.

The investigators would create a new tool able to perform a women's triage, and to detect which of them have to see an anesthesist during a face-to-face consultation and which of them could do without it.

Those types of pre-anesthesic evaluations have already been tested in other countries. A controlled randomized study, executed in Australia between 2012 and 2013, showed the feasibility of a non "in-person" evaluation (by phone, with the aid of an informatic tool and a anesthesist proofreading). Considering these results, the investigators think that it is possible to transpose this type of evaluation to the obstetrical field.

Investigators' study will be about the monocentric analysis of a pre-anesthesic numerical evaluation with the aid of a questionnaire, vouched for by an experts committee specialized in obstetrical anesthesia.

Ultimately, investigators' ambition is to carry out a national multicentric study to analyze this tool on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Major women profiting of a planned pre-anesthesic consultation
* Women who received complete information on research management and who didn't refuse to her participation and her data use.

Exclusion Criteria:

* Participation refusal
* Women without liberty because of a legal or administrative decision
* Women who benefit of psychiatric cares
* Underage women
* Women with legal protection (ex : guardianship)
* Women who can't express their consent
* Language barrier
* Precarious social situation
* Medical pregnancy interruption, foetal death in utero

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is the women who benefit from a classical pre-anesthesic consultation in maternity hospital of Nancy.
Sampling Method: Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Validated Pre-Anesthesic Numerical Evaluation questionnaire | Before enrollment of first pregnant women and during pre-anesthetic consultation of the 8th month.
  Conception of a new and numerical tool for the obstetrical pre-anesthesic evaluation of pregnant women during their pregnancy follow-up. This conception will contain, first, the creation of the questionnaire and then the assessment of the questionnaire's effectiveness in a monocentric study.

SECONDARY OUTCOMES:
Elaborate and validate the first version of Pre-Anesthesic Numerical Evaluation questionnaire | Before enrollment of first pregnant women
  Using the French Health Authority's method published in 2010 : " Recommendations by formalized consensus", validation of the questionnaire with the aid of an experts committee specialized in obstetrical anesthesia.
Validate the first version of Pre-Anesthesia Numerical Evaluation within the population of pregnant women of Maternity Hospital of Nancy (France) | During pre-anesthetic consultation of the 8th month
  Compare the 8th month pre-anesthesic evaluation realized during the classical pre-anesthesic consultation in comparison with the new tool of pre-anesthesic numerical evaluation. The comparison will be proceed thanks to a composite endpoint including birth mode : vaginal delivery or caesarean.
Validate the first version of Pre-Anesthesia Numerical Evaluation within the population of pregnant women of Maternity Hospital of Nancy (France) | During pre-anesthetic consultation of the 8th month
  Compare the 8th month pre-anesthesic evaluation realized during the classical pre-anesthesic consultation in comparison with the new tool of pre-anesthesic numerical evaluation. The comparison will be proceed thanks to a composite endpoint including American Society of Anesthesiologists (ASA) score : 1 (better outcome), 2, 3, 4 or 5.
Validate the first version of Pre-Anesthesia Numerical Evaluation within the population of pregnant women of Maternity Hospital of Nancy (France) | During pre-anesthetic consultation of the 8th month
  Compare the 8th month pre-anesthesic evaluation realized during the classical pre-anesthesic consultation in comparison with the new tool of pre-anesthesic numerical evaluation. The comparison will be proceed thanks to a composite endpoint including existence of bleeding diathesis : Yes or No.
Validate the first version of Pre-Anesthesia Numerical Evaluation within the population of pregnant women of Maternity Hospital of Nancy (France) | During pre-anesthetic consultation of the 8th month
  Compare the 8th month pre-anesthesic evaluation realized during the classical pre-anesthesic consultation in comparison with the new tool of pre-anesthesic numerical evaluation. The comparison will be proceed thanks to a composite endpoint including existence of non-physiologic pregnancy : physiologic pregnancy or non-physiologic pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Bouaziz, MD, PhD, Principal Investigator — Central Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No